CLINICAL TRIAL: NCT02999750
Title: EXACT: EXtendedAnalysis for Cancer Treatment A Prospective Investigator-initiated Translational Study Evaluating Individualized Treatment Regiments Based on Respective Biomarker Analyses for Refractory Cancer Patients
Brief Title: EXtendedAnalysis for Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerald Prager, Univ. Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXACT
Record Dates: First submitted 2016-12-07; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- individual therapy (Other): individual therapy
  Interventions: Other: individual therapy

INTERVENTIONS:
Other: individual therapy — Patient will be treated with individual therapy.

SUMMARY:
The purpose of this study is to prospectively validate treatment benefit of an individualized treatment concept based on molecular profiling (MP) from paraffin-embedded tumor tissue sections obtained before the start of treatment (real time biopsy).

DETAILED DESCRIPTION:
The treatment concept will be considered to be of clinical benefit for the individual patient if a progression-free survival (PFS) ratio (PFS on MP-based therapy / best PFS achieved by prior therapy) will be > 1.0 thus generating a patient cohort with this very property. Thereby, the null hypothesis (that ≤ 40 % of this patient population would have a PFS ratio of > 1.0) will be evaluated with each patient being his own control. For tumor types with high numbers of patients per cohort, the overall response rate (ORR) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients of >19 years with advanced cancer fulfilling the criteria of having:

* an advanced malignancy with metastatic spread refractory to conventional treatment
* a life expectancy of >4 months,
* the possibility to access and biopsy tumour material within 4 weeks before onset of individualized treatment,
* a malignancy amenable to further treatment options with either cytotoxic drugs, tyrosine kinase inhibitors, monoclonal antibodies or related molecules with anti-proliferative potential to cancer cells, as assessed by the ex vivo analysis and a likelihood of treatment response according to the mathematical model (all outlined in detail above),
* agreed to participate by their signature on an informed consent form are eligible.

Exclusion Criteria:

* Presence of further treatment options, as defined by NCCN guidelines which are available in Austria representing a possible further treatment-related response by conventional therapies according to generally accepted medical evidence.
* No fresh and viable tumor material available.
* Current use of therapeutic warfarin.
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) Grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs.
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History of other malignancy. Subjects who have been disease-free for 5 years or those with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Uncontrolled medical conditions (i.e, diabetes mellitus, hypertension, etc), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol)
* unwillingness or inability to follow the procedures required in the protocol.
* pregnant or lactating females.
* History of alcohol or drug abuse within 6 months prior to screening.
* No informed consent available.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Use of real time biopsy to establish an individual molecular profile by using next generation sequencing | 2 years
  pathological examination (includes genetic and target expression profiling, and drug sensitivity screening) to rank treatment options and the potential correlation between treatment response and progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- AKH Vienna, Vienna, Vienna, Austria